CLINICAL TRIAL: NCT00748930
Title: The Canadian ATTRACT Follow-up Program
Brief Title: The Canadian Follow-up Program for the ATTRACT Study (P04868)(TERMINATED)
Status: Terminated | Type: Observational
Why Stopped: Challenging data collection
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04868
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects previously enrolled in the ATTRACT trial from three Canadian sites.
  Interventions: Other: Retrospective Chart Review and Data collection

INTERVENTIONS:
Other: Retrospective Chart Review and Data collection — Retrospective Chart Review and Data collection

SUMMARY:
This is a Phase 4, retrospective chart review of subjects that participated in the ATTRACT study. Site investigators will conduct a chart review and complete a data collection form. The purpose of this study is to describe the treatment used and clinical outcomes of these subjects following completion of the ATTRACT trial up until their most recent assessment by the treating physicians.

DETAILED DESCRIPTION:
Subjects were selected for this study using a non-probability sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been enrolled in the two year follow-up phase of ATTRACT and have continued treatment with the site investigator
* Signature of informed consent.

Exclusion Criteria:

* Not specified in the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects previously enrolled in the ATTRACT trial from three Canadian sites.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To describe the treatment used after completion of the ATTRACT trial in patients enrolled as subjects in the ATTRACT trial from Canadian sites. | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
To describe the long-term therapeutic response as measured by the ACR status in patients enrolled as subjects in the ATTRACT trial from Canadian sites. | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.

SECONDARY OUTCOMES:
To describe the long term safety of infliximab in patients enrolled as subjects in the ATTRACT trial from Canadian sites. | Adverse events will be recorded only for the period after completion of the ATTRACT follow-up.
Disease Activity Score (DAS) | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Morning stiffness | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Swollen joint count | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Tender joint count | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Rheumatoid factor (RF) presence | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
C-reactive Protein (CRP) values | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Erythrocyte Sedimentation Rate (ESR) values | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Annualized X-ray Progression before and after infliximab | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Health Assessment Questionnaire | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Pain Score | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Patient Global Assessment of Disease Status | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Physician Global Assessment of Disease Status | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.
Healthcare Utilization | There are no study specific visits, or patient assessments. Measurements to be recorded for the following time points: Prior to enrollment in ATTRACT, at completion of ATTRACT and for a minimum of three time points after completion of ATTRACT follow-up.